CLINICAL TRIAL: NCT04785092
Title: All Autologous Cartilage Regeneration in the Treatment of the Knee Cartilage Defects: Pilot Study
Brief Title: All Autologous Cartilage Regeneration in the Treatment of the Knee Cartilage Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AACR
Record Dates: First submitted 2021-02-15; First posted 2021-03-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cartilage Damage; Cartilage Disease
Keywords: cartilage; cartilage defect; articular cartilage repair; All Autologous Cartilage Repair; Autologous Chondrocyte Transplantation
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment - All Autologous Cartilage Regeneration (Experimental)
  Interventions: Procedure: All Autologous Cartilage Regeneration

INTERVENTIONS:
Procedure: All Autologous Cartilage Regeneration — All patients will undergo firstly to a blood sampling and then to the arthroscopic debridement of the damage cartilage and subsequently will be harvested the surrounding healthy cartilage The harvested and healthy cartilage will shredded directly in situ with a shaver. This cartilage will then mixed with the patient's own Platelet Concentrate and may be injected directly into the cartilage defect. The Platelet Concentrate stimulates the healing of the cartilage most effectively. At the same time, the Platelet Concentrate will also used to produce autologous fibrin glue, which can be used to fix the applied cartilage chip / Platelet Concentrate product quickly and safely in the damaged cartilage.
  Other Names: Autologous cartilage transplantation

SUMMARY:
The cartilage articular defects of the knee are extremely disabling lesions and represent one of the predisposition causes to the development of articular arthrosis.

When clinical symptoms are present, exist the indication to treat the patient surgically, to this end, several surgical techniques could be performed, as the microfractures, osteochondral transplantation (OCT) or chondrocytes autologous transplantation (ACT).

The aim of this pilot study is to evaluate the clinical performance of a modified version of the ACT technique, the All Autologous Cartilage Repair technique (AACR). A one-step technique in which the healthy cartilage harvested is fragmented directly in situ and then mixed with the autologous platelet concentrate and directly injected in the cartilage defect.. This lead to a less invasive surgery and cost-effective procedure.

The performance will be evaluated through the evaluation of clinical results and complications after surgery other than the evaluation of the quality of the cartilage tissue repaired.

DETAILED DESCRIPTION:
The aim of the Pilot Study is to describe the clinical performance of the AACR technique in the treatment of the cartilage defects in terms of complications after surgery, quality of the repaired cartilage tissue and clinical results with regard to pain and function of the treated knee.

The quality of the repaired cartilage tissue will be evaluate through MRI and clinical outcomes by the Patient Reported Outcome Measures (PROMs).

All patients will undergo to a blood sample (used to product the patient's own platelet concentrate) and an arthroscopic procedure to debride degenerated cartilage tissue and to the harvesting of the surrounding healthy cartilage. The fragmented healthy cartilage will mixed with the platelet concentrate (PC) and injected directly into the cartilage defect to fill it. The platelet concentrate stimulates the healing of the cartilage most actively.

Before and after surgical treatment all patient will undergo to a follow-up visits after 6, 12 and 24 months. MRI will be performed at pre-surgery visit and at the 12 and 24 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Singular symptomatic chondral lesion classified as ICRS III or IV at the femoral condyle with less than 3 mm bone damage under the subchondral plate;
* Lesion between 1 and 8 cm2;
* BMI ≤ 34;
* Ability and will to actively participate in a strict rehabilitation protocol and follow-up.

Exclusion Criteria:

* Previous cartilage operation on the injured knee
* Additional grade III or IV lesion on the same knee
* Previous arthroscopic treatments that affect the AACR technique
* Ligamentous/patellofemoral instability/malposition, varus or valgus malposition ≤3° which cannot be treated/corrected simultaneously
* Previous tendon repair, ligament reconstruction or realignment within the last 6 months
* Any known human immunodeficiency virus, hepatitis, syphilis, malignancy or uncontrolled diabetes
* Uncooperative patients who disregard or cannot follow instructions, including those who abuse drugs and/or alcohol
* Participation in a clinical drug or medical device trial that clinically interferes with the present observational study
* Inability to follow procedures (i.e. dementia)
* Inability to give consent
* No understanding of German language
* Pregnant or lactating women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Change in knee functionality assessed by KOOS | (before treatment, 6, 12 and 24 months postoperative
  The primary clinical outcome is the change in knee functionality assessed by the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire over 2 years (before treatment, at baseline, versus 6, 12 and 24 months postoperative). The KOOS is a Patient Reported Outcome Measure (PROM) designed to asses patient-relevant outcomes following knee injury.
  It is a self-completion questionnaire with a 1-week-recall-period with 42 items and 5 subscales (pain, symptoms, activities of daily life, sport and leisure, quality of life associated with the knee joint). Each question has five answering options, scored with a numerical value of 0 - 4. In average, it takes 10 minutes to complete. The calculation of the respective sub-score is done by adding up the marked items of the relevant subscales. These numerical values are then converted into a scale value between 0 (extreme knee problems) and 100 (free of knee joint complaints).

SECONDARY OUTCOMES:
Quality of cartilage repair tissue MRI evaluation | 12 and 24 months
  The quality of cartilage repair tissue will be assessed with the Magnetic Resonance Observation of Cartilage Repair Tissue (MOCART). The MOCART score is the variable of primary interest because it allows both the evaluation of cartilage repair tissue and the surrounding structures. The MOCART score is based on nine variables measured on a standard MRI and added up to a score, ranging from 0 to 100, where 100 represents the best score and a score of 0 represents the worst score.
Difference between baseline and follow-up visits of the physical examination | Baseline, 6, 12 and 24 months
  The physical examination will evaluate the knee swelling, dynamic and static alignment.
Marx activity rating scale (MARS) | Baseline, 6, 12 and 24 months
  is patient-administered and takes only 1 minute to complete. It includes 4 items that assess the frequency of running, cutting, decelerating, and pivoting based on the subjects "healthiest and most active state in the past year." Each question has five answering options, scored with a numerical value of 0 - 4. The score of all items is summed up for the total score, which ranges from 0 (lowest physical or sporting activity) to 16 (highest physical or sporting activity).
Numeric Rating Scale (NRS) for pain | Baseline, 6, 12 and 24 months
  is a single item question about the average pain on ordinary days with average physical activity, where numerical answers are anchored by 0 (no pain) and 10 (worst possible pain)
Baseline quality of cartilage repair tissue MRI evaluation | baseline
  The AMADEUS (Area Measurement And DEpth & Underlying Structures) scoring system includes the three most important different parameters that describe a focal chondral or osteochondral defect prior to possible cartilage repair surgery: (1) the cartilage defect area, which is measured ("area measurement"); (2) the cartilage defect morphology/depth ("depth"); and (3) the underlying structures with presence of adjacent osseous defects/subchondral cysts and bone marrow edema-like lesions (BME) ("under- lying structures"). In addition to the resulting AMADEUS code, sub-scores were defined for each feature, which sum up to a total score of 100 (no osteochondral defect) to 0 (worst score).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Na Y, Shi Y, Liu W, Jia Y, Kong L, Zhang T, Han C, Ren Y. Is implantation of autologous chondrocytes superior to microfracture for articular-cartilage defects of the knee? A systematic review of 5-year follow-up data. Int J Surg. 2019 Aug;68:56-62. doi: 10.1016/j.ijsu.2019.06.007. Epub 2019 Jun 18. PMID 31220632
- [Background] Brittberg M, Lindahl A, Nilsson A, Ohlsson C, Isaksson O, Peterson L. Treatment of deep cartilage defects in the knee with autologous chondrocyte transplantation. N Engl J Med. 1994 Oct 6;331(14):889-95. doi: 10.1056/NEJM199410063311401. PMID 8078550
- [Background] Massen FK, Inauen CR, Harder LP, Runer A, Preiss S, Salzmann GM. One-Step Autologous Minced Cartilage Procedure for the Treatment of Knee Joint Chondral and Osteochondral Lesions: A Series of 27 Patients With 2-Year Follow-up. Orthop J Sports Med. 2019 Jun 13;7(6):2325967119853773. doi: 10.1177/2325967119853773. eCollection 2019 Jun. PMID 31223628
- [Background] Brittberg M, Peterson L, Sjogren-Jansson E, Tallheden T, Lindahl A. Articular cartilage engineering with autologous chondrocyte transplantation. A review of recent developments. J Bone Joint Surg Am. 2003;85-A Suppl 3:109-15. doi: 10.2106/00004623-200300003-00017. No abstract available. PMID 12925617